CLINICAL TRIAL: NCT01957111
Title: Metabolomics of Insomnia-Related Hyperarousal
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MISP-50802
Record Dates: First submitted 2013-09-17; First posted 2013-10-08 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Individuals with insomnia
- Good sleepers

SUMMARY:
Individuals with insomnia have been shown to have higher overall metabolic rates compared to good sleepers, but it is not known which metabolic processes are involved. The goal of this study is to compare a wide array of metabolic processes in 15 people with insomnia and 15 good sleepers. We hypothesize that there will be distinct metabolic processes that are functioning differently in those with insomnia.

ELIGIBILITY:
Inclusion Criteria:

Criteria for primary insomnia:

* subjective complaint of difficulty initiating or maintaining sleep, waking up too early or nonrestorative sleep
* daytime consequences as a result of the poor sleep
* duration of at least 1 month
* sleep disturbance is not secondary to a medical or psychiatric condition

Criteria for good sleepers:

-subjective report of consistent good sleep

Exclusion Criteria:

* significant medical or psychiatric illness
* diagnosis of a sleep disorder other than insomnia
* women who have been pregnant or lactating in the past 6 months
* non-fluency in spoken or written English
* Current shift work defined as working during the evening or night shift
* Current use of medications that affect sleep
* BMI >27

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals with primary insomnia (n=15) and matched good sleepers (n=15)
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gehrman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Gehrman P, Sengupta A, Harders E, Ubeydullah E, Pack AI, Weljie A. Altered diurnal states in insomnia reflect peripheral hyperarousal and metabolic desynchrony: a preliminary study. Sleep. 2018 May 1;41(5):zsy043. doi: 10.1093/sleep/zsy043. PMID 29522222

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the general community and consisted of a group of with chronic insomnia disorder and age- and sex-matched good sleepers.
Groups:
- Individuals With Insomnia: Participants with insomnia met the following Research Diagnostic Criteria for primary insomnia: subjective complaint of difficulty initiating or maintaining sleep, waking up too early or nonrestorative sleep, daytime consequences as a result of the poor sleep, duration of at least 1 month, sleep disturbance is not secondary to a medical or psychiatric condition based or the effects of a substance, as determined by clinical history. In order to exclude individuals with mild insomnia, insomnia had to occur on 3 or more nights per week for three months or longer. A 30-minute criterion was used such that subjects had to report taking 30 minutes or longer to fall asleep and/or spend 30 minutes awake during the night.
- Good Sleepers: To be considered a good sleeper, participants had to report that they did not have difficulty falling asleep or staying asleep. A 15-minute criterion was used such that subjects had to report taking 15 minutes or less to fall asleep and spend 15 minutes or less awake during the night.
Period: Overall Study
Arm/Group | Individuals With Insomnia | Good Sleepers
Started | 16 | 16
Completed | 15 | 15
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individuals With Insomnia | Good Sleepers | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (7.9) | 36.0 (7.5) | 36.5 (7.7)
Gender [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 12 | 14 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Metabolites Elevated Relative to the Other Group.
Description: Metabolomics analysis of blood samples were carried out using Spectroscopy. This approach allows for rapid, unbiased and quantitative metabolic profiles ('fingerprints) to be acquired. A total of 70 metabolites were measured and compared between individuals with insomnia and good sleepers.
Time Frame: 48 hours
Measure: Number; unit: Number of metabolites elevated
Arm/Group | Individuals With Insomnia | Good Sleepers
Number analyzed (Participants) | 15 | 15
Number of metabolites elevated | 13 | 9

2. Secondary Outcome: Sleep Efficiency Percentage on Overnight Sleep Study
Description: Participants will have their sleep measured with polysomnography for one night. The sleep of individuals with insomnia will be compared to that of good sleepers. Sleep quality is defined as sleep efficiency, which is calculated at total sleep time / total time spent in bed x 100. It indicates the % of time spent asleep while in bed.
Time Frame: 1 night
Measure: Mean (Standard Deviation); unit: % sleep efficiency
Arm/Group | Individuals With Insomnia | Good Sleepers
Number analyzed (Participants) | 15 | 15
% sleep efficiency | 75.8 (14.6) | 80.7 (9.8)

ADVERSE EVENTS:
Arm/Group | Individuals With Insomnia | Good Sleepers
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No